CLINICAL TRIAL: NCT05203978
Title: Virtual Reality Colonoscopy : a Study From Nancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Baptiste CHEVAUX, Hospital practitioner, Central Hospital, Nancy, France
Other Study IDs: 2021PI080
Record Dates: First submitted 2021-11-29; First posted 2022-01-24 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Neoplasms; Colorectal Polyp
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Virtual reality colonoscopy: using virtual reality with glasses and sound no anaesthesia
  Interventions: Procedure: colonoscopy
- General anaesthesia colonoscopy: gold standard
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: colonoscopy — Colonoscopy

SUMMARY:
Colonoscopy is an exam which can be responsible for pain and discomfort for the patient.

Therefore colonoscopy is performed most of the time under general anaesthesia. Moreover, drug-induced sedation comes with adverse effects especially among fragile patients.

Besides, monitoring patients during and after sedation is both logistically demanding and costly.

Virtual reality offers immersive and three dimensional experiences that distract the attention and might improve patients comfort.

The aim of the study is to investigate the use of virtual reality during colonoscopy versus general anaesthesia.

DETAILED DESCRIPTION:
The study is based on a home made questionnaires completed by the operator and the patient before and after the colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* patient needed planned colonoscopy
* able to fill in questionnaires in French

Exclusion Criteria:

* visual or auditor impairments
* dementia patient
* limited French language skills
* diagnosis of balance disorders or epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient needed planned colonoscopy and able to fill in questionnaires in French
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Complete colonoscopy defined by caecum intubation (binary criterion : yes or no) | baseline
  found of the report

SECONDARY OUTCOMES:
Pain evaluated by Numeric Rating Scale during the procedure (0 no pain and 10 highest imaginable pain) | baseline
  asked on the questionnaire
Anxiety evaluated by the validated score State Trait Anxiety Inventory ranging from 20 (absence of anxiety) to 80 (highest anxiety) | baseline
  asked on the questionnaire
Comfort evaluated by Gloucester Comfort Scale between 1 comfortable and 5 severe discomfort | baseline
  asked on the questionnaire
Satisfaction evaluated on scale of willingness to return (0 no willing at all to 10 definitively willing) | baseline
  asked on the questionnaire
Polyp removal (binary criterion : yes or no) | baseline
  found on the report